CLINICAL TRIAL: NCT06352684
Title: Multi-Reader Multi-Case, Retrospective Study to Evaluate Effectiveness of CadAI-B for Breast
Status: Active, not recruiting | Type: Observational
Sponsor: BeamWorks Inc. (Industry)
Collaborators: Severance Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: DP0001-SEV-CAB-II; RS-2023-00227526 (Other Grant/Funding Number: Korea Ministry of Science and ICT)
Record Dates: First submitted 2024-04-02; First posted 2024-04-08 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (3):
- Cancer group: confirmed as a breast cancer (DCIS or invasive cancer) through the subsequent biopsy conducted within following 1 year of the ultrasound exam.
  Interventions: Device: CadAI-B for Breast
- Benign group: Either confirmed as a benign through the subsequent biopsy conducted within following 1 year of the ultrasound exam or showing stability on more than 2 years of imaging follow-up after initial diagnosis
  Interventions: Device: CadAI-B for Breast
- Normal group: Interpreted as BI-RADS 1 (Negative) with no cancers on the ultrasound exam
  Interventions: Device: CadAI-B for Breast

INTERVENTIONS:
Device: CadAI-B for Breast — CadAI-B for Breast is designed to assist healthcare professionals in lesion detection and differential diagnosis during breast US examinations.

SUMMARY:
The purpose of this study is to evaluate the effectiveness of lesion detection and diagnosis-aiding software (CadAI-B for Breast) during ultrasound (US) examination

DETAILED DESCRIPTION:
CadAI-B for Breast is a real-time AI diagnosis system designed to assist healthcare professionals in lesion detection and differential diagnosis during breast US examinations. The primary objective of the study is to evaluate the effectiveness of CadAI-B in the assistance of detection and diagnosis of breast cancer by comparing the clinical performance of physicians before and after using CadAI-B in their ultrasound reading. The secondary objective of this study is to evaluate the sensitivity and specificity using CadAI-B for US examinations.

ELIGIBILITY:
Inclusion Criteria:

* Women who underwent breast US examination
* Women with breast cancer (DCIS or invasive cancer) diagnosed via biopsy
* Women who had been followed for more than 2 years after initial US examination

Exclusion Criteria:

* women who had breast implants
* women who had US images containing artifacts affecting the review of images

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Mainly recruited from a tertiary hospital but no limitation of enrollment
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2023-11-24 (Actual); Primary Completion 2025-01-14 (Estimated); Study Completion 2025-01-14 (Estimated)

PRIMARY OUTCOMES:
Area Under the LROC Curve | 6 weeks
  The area under the LROC curve (AUC_LROC) on the diagnosis of suspicious lesions was computed and compared between the aided and unaided sessions.

SECONDARY OUTCOMES:
Lesion detection sensitivity and specificity | 6 weeks
  The mean sensitivity and specificity of 15 readers were calculated and compared between the aided and unaided sessions.

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University Severance Hospital, Seoul, South Korea